CLINICAL TRIAL: NCT02379455
Title: Cooperation for Improved Pharmacotherapy in Home-dwelling Elderly People Receiving Polypharmacy - The COOP Study
Acronym: COOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Torgeir Bruun Wyller, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 222033/H10
Record Dates: First submitted 2015-02-27; First posted 2015-03-05 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Drug Usage
Keywords: Polypharmacy; Geriatrics; Elderly; Drug review

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive drug review (Experimental)
  Interventions: Other: Comprehensive drug review
- Control group (No Intervention): Follow-up by family physician "as usual".

INTERVENTIONS:
Other: Comprehensive drug review — 1) Geriatric assessment including medical history, physical examination, supplementary tests. The geriatric work-up will be aimed at evaluating whether current medications are indicated, whether the relevant conditions are satisfactorily compensated, whether the dosages are appropriate, whether the patient has symptoms that may in reality be adverse drug effects, and whether drug-drug interactions or drug-disease interactions are likely to occur. 2) Conference with common drug review. The project physician and the family physician will discuss the patient's drug list systematically. 3) Individualized clinical follow-up depending on the medication changes that have been done.
  Arms: Comprehensive drug review

SUMMARY:
Polypharmacy increases the risk of adverse drug effects, interactions and other drug-related problems, and several studies indicate that inappropriate drug use is a major reason for poor health and impaired function in the elderly. A majority of interventions for improvement of drug treatment in the elderly have been evaluated by the use of surrogate outcomes such as drug-related problems, number of prescribed drugs or prevalence of potentially inappropriate prescriptions - and it is so far unclear whether such interventions can result in clinical significant improvements. The primary objective of this trial is therefore to evaluate the effect upon patients, relatives and local health care service of a structured cooperation between a hospital-based geriatrician and family physicians on complex drug regimens in home-dwelling frail elderly patients.

DETAILED DESCRIPTION:
This is a 24 weeks cluster randomized, single-blinded, controlled trial. Family physicians will be invited to participate in the project with patients from their lists, and can participate with 1-5 patients each. The investigators will carry out cluster randomization on physician level instead of individual randomization on patient level.

The investigators suppose that such a comprehensive clinical evaluation and drug review that they will test, is most relevant for patients with relatively pronounced polypharmacy. It has previously been shown that conventionally used limits for polypharmacy, e.g. five drugs used regularly, identifies many patients without particular complex health states and without drug related problems. The investigators will therefore limit this project to patients using seven regular drugs or more, in order to increase the likelihood that they may benefit from a drug review.

A major challenge when studying complex interventions is to describe the intervention with sufficient precision as to facilitate replication. Our main strategy for this will be to compensate for the necessary degree of pragmatism in the interventional approach with a detailed description of the interventions that were in fact carried out, in particular changes in the drug regimens of the individual patients.

The intervention will consist of three main parts:

1. Geriatric assessment: The patients will be seen by a physician trained in geriatric medicine. The physician will carry out a medical history and a physical examination, and relevant blood analyses and other supplementary test will be ordered if not already available. The geriatric work-up will be aimed at evaluating whether current medications are indicated, whether the relevant conditions are satisfactorily compensated, whether the dosages are appropriate, whether the patient has symptoms that may in reality be adverse drug effects, and whether drug-drug interactions or drug-disease interactions are likely to occur. Published tools like the START (Screening Tool of Older Persons' Prescriptions) criteria, Screening Tool to Alert doctors to Right Treatment (STOPP) criteria and The Norwegian General Practice (NORGEP) criteria will be used.
2. Conference with common drug review: The main purpose of this conference is to combine the competence of the geriatrician and that of the family physician in a focused drug review. The two physicians will discuss the patient's drug list systematically. The geriatrician may suggest changes in the drug regimen, but the family physician retains the medical responsibility for the patient and is in charge of all ordinations and medication changes.
3. Clinical follow-up: Depending on medication changes that have been done, the two physicians will arrange the necessary follow-up within the project period.

The investigators will assess the outcomes at 16 and 24 weeks, counted from baseline, and will also assess baseline values for the outcomes in order to adjust for potential inequalities.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be on the list of one of the family physicians participating in the study
* Home dwelling (not permanently institutionalised)
* Medications administered by the home nursing service
* Polypharmacy defined as the use of at least seven different systemic medications taken regularly
* Informed consent by the patient or a close relative

Exclusion Criteria:

* Patient or relative denies inclusion
* The family physician does not want the particular patient to participate
* Moderate/severe dementia (Clinical Dementia Rating Scale score > 1) and contact with the closest proxy less than once every other week.
* The patient does not speak/understand Norwegian
* Expected to become permanently institutionalised within six months
* Life expectancy < six months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life as measured with 15D | 16 weeks

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 16 weeks
Short Physical Performance Battery (SPPB) | 24 weeks
Gait speed | 16 weeks
Gait speed | 24 weeks
Hand grip strength | 16 weeks
Hand grip strength | 24 weeks
Functional Independence Measure (FIM) | 16 weeks
Functional Independence Measure (FIM) | 24 weeks
Trail making test A and B | 16 weeks
Trail making test A and B | 24 weeks
Digit Span | 16 weeks
Digit Span | 24 weeks
Five Digits Test | 16 weeks
Five Digits Test | 24 weeks
Medication Appropriateness Index (MAI) | 16 weeks
Medication Appropriateness Index (MAI) | 24 weeks
Assessment of Underutilization (AOU) | 16 weeks
Assessment of Underutilization (AOU) | 24 weeks
Number of falls | During the first 16 weeks after baseline
  Recorded with the aid of diaries kept by patients/caregivers
Number of falls | During the first 24 weeks after baseline
  Recorded with the aid of diaries kept by patients/caregivers
Orthostatic blood pressure | 16 weeks
Orthostatic blood pressure | 24 weeks
Changes in body weight | 16 weeks
Changes in body weight | 24 weeks
Relative Stress Scale | 16 weeks
Relative Stress Scale | 24 weeks
Number of hospital admissions (with reasons) | During the first 16 weeks from baseline
Number of hospital admissions (with reasons) | During the first 24 weeks from baseline
Number of days in own home (in contrast to being in hospital or nursing home) | During the first 16 weeks from baseline
Number of days in own home (in contrast to being in hospital or nursing home) | During the first 24 weeks from baseline
Admission to permanent institutional care | 16 weeks
Admission to permanent institutional care | 24 weeks
Current use of home nursing service | 16 weeks
Current use of home nursing service | 24 weeks
Mortality | 16 weeks
Mortality | 24 weeks
Health-related quality of life as measured with 15D | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir B Wyller, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Dept. of Geriatric Medicine, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Veddeng S, Madland H, Molden E, Wyller TB, Romskaug R. Association between statin use and physical performance in home-dwelling older patients receiving polypharmacy: cross-sectional study. BMC Geriatr. 2022 Mar 23;22(1):242. doi: 10.1186/s12877-022-02942-7. PMID 35321652
- [Derived] Romskaug R, Skovlund E, Straand J, Molden E, Kersten H, Pitkala KH, Lundqvist C, Wyller TB. Effect of Clinical Geriatric Assessments and Collaborative Medication Reviews by Geriatrician and Family Physician for Improving Health-Related Quality of Life in Home-Dwelling Older Patients Receiving Polypharmacy: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2020 Feb 1;180(2):181-189. doi: 10.1001/jamainternmed.2019.5096. PMID 31617562
- [Derived] Romskaug R, Molden E, Straand J, Kersten H, Skovlund E, Pitkala KH, Wyller TB. Cooperation between geriatricians and general practitioners for improved pharmacotherapy in home-dwelling elderly people receiving polypharmacy - the COOP Study: study protocol for a cluster randomised controlled trial. Trials. 2017 Apr 4;18(1):158. doi: 10.1186/s13063-017-1900-0. PMID 28372591